

## NON-INTERVENTIONAL (NI) STUDY PROTOCOL

## **Study Information**

| Title | Effect of Trumenba on Gonococcal infections in adolescents and young adults in the United States: A retrospective cohort study |
|---|---|
| Protocol number | B1971066 |
| Protocol version identifier | 1.0 |
| Date | 18 April 2023 |
| Medicinal product | Trumenba |
| Research question and objectives | To examine the effect of Trumenba on gonococcal infection in adolescents and young adults in the United States using a claims database. |
| Author | PPD (Pfizer): PPD (Pfizer): PPD PPD (Pfizer): PPD PPD (Pfizer): PPD |

This document contains confidential information belonging to Pfizer. Except as otherwise agreed to in writing, by accepting or reviewing this document, you agree to hold this information in confidence and not copy or disclose it to others (except where required by applicable law) or use it for unauthorized purposes. In the event of any actual or suspected breach of this obligation, Pfizer must be promptly notified.

## 1. TABLE OF CONTENTS

| 1. TABLE OF CONTENTS | 2 |
|---|---|
| 2. LIST OF ABBREVIATIONS | 4 |
| 3. RESPONSIBLE PARTIES | 6 |
| 4. ABSTRACT | 7 |
| 5. AMENDMENTS AND UPDATES | 8 |
| 6. MILESTONES | 9 |
| 7. RATIONALE AND BACKGROUND | 10 |
| 8. RESEARCH QUESTION AND OBJECTIVES | 11 |
| 8.1. Objectives | 11 |
| 8.1.1. Primary Objective | 11 |
| 8.1.2. Secondary Objectives | 11 |
| 8.1.3. Exploratory Objectives | 11 |
| 9. RESEARCH METHODS | 11 |
| 9.1. Study Design | 11 |
| 9.2. Setting | 12 |
| 9.2.1. Inclusion Criteria | 12 |
| 9.2.2. Exclusion Criteria | 12 |
| 9.3. Variables | 12 |
| 9.4. Data Sources | 17 |
| 9.5. Study Size | 17 |
| 9.6. Data Management | 18 |
| 9.7. Data Analysis | 18 |
| 9.8. Quality Control | 18 |
| 9.9. Strengths and Limitations of the Research Methods | 19 |
| 9.10. Other Aspects | 19 |
| 10. PROTECTION OF HUMAN SUBJECTS | 19 |
| 10.1. Patient Information. | 19 |
| 10.2. Patient Consent | 19 |
| 10.3. Institutional Review Board (IRB)/Independent Ethics Committee (IEC) | 19 |
| 10.4. Ethical Conduct of the Study | 20 |

| 11. MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS | 20 |
|------------------------------------------------------------------|----|
| 12. PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS | |
| 13. REFERENCES | 21 |
| 14. LIST OF TABLES | 22 |
| 15. LIST OF FIGURES | 22 |
| ANNEX 1. LIST OF STAND ALONE DOCUMENTS | 22 |

## 2. LIST OF ABBREVIATIONS

| Abbreviation | Definition |
|---|---|
| 4CMenB | bexsero vaccine |
| CIOMS | International Ethical Guidelines for Epidemiological<br>Research issued by the Council for International<br>Organizations of Medical Sciences |
| CFR | Code of Federal Regulations |
| CPT | current procedural terminology |
| EMA | European Medicines Agency |
| ENCePP | European Network of Centres for Pharmacoepidemiology and Pharmacovigilance |
| FDA | Food and Drug Administration |
| fHBP | factor H binding protein |
| GEP | Good Epidemiological Practice |
| GPP | Good Pharmacoepidemiology Practices |
| HRs | hazard ratios |
| HIPAA | Health Insurance Portability and Accountability Act |
| HIV | human immunodeficieny virus |
| ICD-10-CM | International Classification of Diseases, 10 <sup>th</sup><br>Revision, Clinical Modification |
| IEA | International Epidemiological Association |
| IEC | Independent Ethics Committee |
| IRB | Institutional Review Board |
| ISPE | International Society for Pharmacoepidemiology |
| ISPOR | Good Outcomes Research Practices issued by the International Society for Pharmacoeconomics and Outcomes Research |
| MenB | Meningococcal Serogroup B |
| MSM | men who have sex with men |
| NDC | National Drug Codes |
| OMV | outer membrane vesicle |
| PASS | Post-Authorization Safety Study |

| Abbreviation | Definition |
|--------------|-----------------------------|
| SAS | statistical analysis system |
| US | United States |
| VE | Vaccine effectiveness |

## 3. RESPONSIBLE PARTIES

## Principal Investigator(s) of the Protocol

| Name, degree(s) | Job Title | Affiliation | Address |
|---|---|---|---|
| Myint Tin Tin Htar | Epidemiology Lead | Pfizer | 23-25 Avenue Docteur<br>Lannelongue 75014<br>Paris, France |
| Mohammad Ali, PhD | Statistician | Pfizer | 500 Arcola Rd<br>Collegeville, PA |
| Angela Quinn, BS | Clincal Scientist | Pfizer | 500 Arcola Rd<br>Collegeville, PA |
| Sarah Jeanette Willis | Director, Vaccines<br>RWE Scientist | Pfizer | Remote, PPD |

## 4. ABSTRACT

Not required.

## 5. AMENDMENTS AND UPDATES

None.

## 6. MILESTONES

| Milestone | Planned date |
|--------------------------|-----------------|
| Start of data collection | 20 April 2023 |
| End of data collection | 30 April 2023 |
| Final study report | 31 October 2023 |

#### 7. RATIONALE AND BACKGROUND

This study is not a Post-Authorization Safety Study (PASS) and is not a commitment to any regulatory authority.

Meningococcal B outer membrane vesicle (OMV) vaccines have been created, developed and used to control outbreaks of meningococcal B diseases in New Zealand, Norway and Cuba. Studies suggested that OMV vaccines could potentially protect against gonococcal infections in New Zealand and Norway.<sup>1</sup>

Recently 4 studies described the effect of Bexsero (4CMenB) on gonococcal infection in adolescents and young adults (2 studies in the United States (US), 1 in Australia and 1 in Italy). The vaccine coverage differed by studies (69% in Australia, 33% in men who have sex with men (MSM) living with human immunodeficiency virus (HIV) in Italy and 1.8% in New York City & Philadelphia. The direct effect of 4CMenB (vaccine effectiveness) ranged from 32 to 74% for 2 full doses and 33 to 71% for at least 1 dose.<sup>2-5</sup>

Abara et al studied the effectiveness of 4CMenB and factor H binding protein (fHbp) vaccines in 2 separate studies using the same methodology in New York and Philadelphia regions for the period of 2016-2018 (the first 2 years of meningococcal serogroup B [MenB] vaccines use in the US). The vaccine coverage was 7.4% and 1.6% for at least one dose for 4CMenB and fHbp vaccines respectively. The effectiveness of 4CMenB was 40% (95% CI 23; 53) for full dose and 26% (95% CI 12; 37) for only 1 dose. The effectiveness of fHbp vaccine was 3% (95%CI: +19; 21).6 6These results were based on data during the period where fHbp had extremely low vaccine coverage (<2%).

The vaccine effectiveness for 4CMenB varied highly according to study types, age of the study population and the vaccine coverage rate. The vaccine coverage had increased to 32% for any MenB vaccines in 2021 while it was 14% and 17% in 2017 and 2018 respectively. The effectiveness of fHbp vaccine observed in Abara et al study could be confirmed in a larger population with higher vaccine coverage. The purpose of the study will be to evaluate the effect of fHbp vaccine in prevention of gonococcal infection among 15-30 years in the US using the claim database.

## 8. RESEARCH QUESTION AND OBJECTIVES

#### 8.1. Objectives

#### 8.1.1. Primary Objective

To examine the effect of at least 1 dose of Trumenba on gonococcal infection in adolescents and young adults of 15-30 years in the US.

## 8.1.2. Secondary Objectives

- 1. To examine the effect of at least 2 doses of Trumenba on gonococcal infection in adolescents and young adults of 15-30 years in the US.
- 2. To examine the effect of at least 1 dose of Trumenba on chlamydial infection in adolescents and young adults of 15-30 years in the US.
- 3. To examine the effect of at least 2 doses of Trumenba on chlamydial infection in adolescents and young adults of 15-30 years in the US.

#### 8.1.3. Exploratory Objectives

- 1. To examine the effect of at least 1 dose of Trumenba on gonococcal infection in adolescents and young adults of 16-23 years in the US.
- 2. To examine the effect of 1 dose of Trumenba on gonococcal infection in adolescents and young adults of 15-30 years in the US at 12 months, 24 months, 36 months and 48 months following the index vaccination.

#### 9. RESEARCH METHODS

#### 9.1. Study Design

This is a retrospective cohort study using health care administrative claims data as described in Section 9.4 Data Sources.

Adolescents and young adults approximately 15 to 30 years of age at their individual time zero (calculated based on birth year) will be identified from administrative claims during 01 January 2016 and 31 December 2021.

The exposure cohort will be the individuals who have received at least 1 dose of Trumenba and at least 1 dose of MenACWY (Menactra®, Menveo®, or MenQuadfi®) prior to the Trumenba vaccination, between 01 January 2016 and 31 December 2021. The index date (zero time) for the exposed cohort is the last date of vaccination, and the cohort will be followed from 14 days after vaccination to the end of the study period (31 December 2022). The individuals in the cohort will be censored by the event of interest, death date (if known), plan disenrollment (if known) or the end of the study period, whichever comes first.

The reference cohort will be those with at least 1 dose of MenACWY vaccine, but no doses of Trumemba during the observation period, received between 01January 2016 and 31 December 2021. The MenACWY-only vaccinated cohort is used as a reference cohort rather than an unvaccinated cohort in order to help control for theoretical differences in health seeking and risk behaviors between vaccinated and unvaccinated individuals. The index date (zero time) of the reference cohort is the last dose of MenACWY and these individuals will be followed from 14 days after zero time until the earliest occurrence of the following: outcome of interest, death date (if known), plan disenrollment (if known) or 31 December 2022 (end of study period).

The outcomes of interest are gonococcal and chlamydial infections and only the first episode within the study period will be considered as event in case of repeated infections.

#### 9.2. Setting

IQVIA PharMetrics® Plus is a longitudinal health plan database of adjudicated medical and pharmacy claims, including patient enrollment data for national and sub-national health plans and self-insured employer groups in the US. Administrative claims and enrollment data available during 01 January 2016 and 31 December 2022 will be used in this study.

#### 9.2.1. Inclusion Criteria

Patient records must meet all of the following inclusion criteria to be eligible for inclusion in the study:

- 1. Individuals of approximately 15-30 years old (using July 1 of birth year) enrolled in a health plan available in PharMetrics Plus database during 01 January 2016 and 31 December 2021.
- 2. Individuals having at least 1 dose of MenACWY during 01 January 2016 and 31 December 2021.

#### 9.2.2. Exclusion Criteria

Patients meeting any of the following criteria will not be included in the study:

Individuals having any dose of Bexsero at any time during 01 January 2016 and 31 December 2021 and prior to the study

Individuals with missing demographic variables or dates of outcome diagnoses or vaccine administration (listed in Section 9.3).

#### 9.3. Variables

In this study, the variables of interest are age, gender, state of residence, date of vaccination and the date of disease diagnosis.

## Table 1. Variable List

| Variable | Role | Operational Definition |
|---|---|---|
| Birth Year | Covariate | Birth year (age to be |
| | | calculated based on July 1 of birth year) |
| Gender | Covariate | Male, Female, Unknown |
| Residence (ZIP code) | Covariate | First 3 digits of the zip |
| Residence (Zii code) | Covariate | code from individuals' |
| | | most recent enrollment |
| M ACMW : 4: | NI | |
| MenACWY vaccination | Non-exposure | Current procedural |
| | | terminology (CPT) codes |
| | | and National Drug |
| | | Codes (NDC) listed |
| | | below |
| Trumemba vaccination | Exposure | CPT and |
| | - | NDCs listed below |
| Gonococcal infection | Primary Outcome | ICD-10-CM codes listed |
| | • | below |
| Chlamydial infection | Reference disease | ICD-10-CM codes listed |
| | Outcome | below |

Table 2. Diagnosis Codes for Identifying Gonococcal Infections

| Code | Туре |
|-------|-----------|
| A540 | ICD-10-CM |
| A5400 | ICD-10-CM |
| A5401 | ICD-10-CM |
| A5402 | ICD-10-CM |
| A5403 | ICD-10-CM |
| A5409 | ICD-10-CM |
| A541 | ICD-10-CM |
| A542 | ICD-10-CM |
| A5421 | ICD-10-CM |
| A5422 | ICD-10-CM |
| A5423 | ICD-10-CM |
| A5424 | ICD-10-CM |
| A5429 | ICD-10-CM |
| A543 | ICD-10-CM |
| A5430 | ICD-10-CM |
| A5431 | ICD-10-CM |
| A5432 | ICD-10-CM |
| A5433 | ICD-10-CM |
| A5439 | ICD-10-CM |
| A544 | ICD-10-CM |
| A5440 | ICD-10-CM |
| A5441 | ICD-10-CM |
| A5442 | ICD-10-CM |
| A5443 | ICD-10-CM |
| A5449 | ICD-10-CM |
| A545 | ICD-10-CM |
| A546 | ICD-10-CM |
| A548 | ICD-10-CM |
| A5481 | ICD-10-CM |
| A5482 | ICD-10-CM |
| A5483 | ICD-10-CM |
| A5484 | ICD-10-CM |
| A5485 | ICD-10-CM |
| A5486 | ICD-10-CM |
| A5489 | ICD-10-CM |
| A549 | ICD-10-CM |

Table 3. Diagnosis Codes for Identifying Chlamydial Infections

| Code | Туре |
|-------|-----------|
| A55 | ICD-10-CM |
| A560 | ICD-10-CM |
| A5600 | ICD-10-CM |
| A5601 | ICD-10-CM |
| A5602 | ICD-10-CM |
| A5609 | ICD-10-CM |
| A561 | ICD-10-CM |
| A5611 | ICD-10-CM |
| A5619 | ICD-10-CM |
| A562 | ICD-10-CM |
| A563 | ICD-10-CM |
| A564 | ICD-10-CM |
| A568 | ICD-10-CM |
| A71 | ICD-10-CM |
| A710 | ICD-10-CM |
| A711 | ICD-10-CM |
| A719 | ICD-10-CM |
| A74 | ICD-10-CM |
| A740 | ICD-10-CM |
| A748 | ICD-10-CM |
| A7481 | ICD-10-CM |
| A7489 | ICD-10-CM |
| A749 | ICD-10-CM |

Table 4. Current Procedural Terminal Codes and National Drug Codes for Identifying MenACWY Vaccination

| Code | Type | Description |
|---------------|------|-----------------------------|
| 90734 | CPT | Menactra/Menveo Vaccination |
| 90619 | CPT | Menquadfi Vaccine |
| 49281-0589-05 | NDC | Menactra Vaccine |
| 46028-0208-01 | NDC | Menveo Vaccine |
| 58160-0955-09 | NDC | Menveo Vaccine |
| 49281-0589-58 | NDC | Menactra Vaccine |
| 49281-0590-58 | NDC | Menquadfi Vaccine |
| 46028-0218-11 | NDC | Menveo Vaccine |
| 58160-0958-01 | NDC | Menveo Vaccine |
| 58160-0959-01 | NDC | Menveo Vaccine |
| 46028-0219-11 | NDC | Menveo Vaccine |
| 54569-5687-01 | NDC | Menactra Vaccine |
| 50090-1890-01 | NDC | Menactra Vaccine |
| 49281-0590-05 | NDC | Menquadfi Vaccine |

Table 5. Current Procedural Terminal Codes and National Drug Codes for Identifying Trumemba (fHbp) Vaccination

| Code | Type | Description |
|---------------|------|----------------------|
| 90621 | CPT | Trumenba Vaccination |
| 00005-0100-01 | NDC | Trumenba Vaccine |
| 00005-0100-02 | NDC | Trumemba Vaccine |
| 00005-0100-05 | NDC | Trumenba Vaccine |
| 00005-0100-10 | NDC | Trumenba Vaccine |

Table 6. Current Procedural Terminal Codes and National Drug Codes for Identifying Bexsero 4CMenB Vaccination

| Code | Type | Description |
|---|---|---|
| 90620 | CPT | Meningococcal recombinant protein and outer membrane vesicle (OMV) vaccine, serogroup B (MenB-4C), 2 dose schedule, for intramuscular use |
| 46028011401 | NDC | Bexsero vaccine |
| 46028011402 | NDC | Bexsero vaccine |
| 46028011411 | NDC | Bexsero vaccine |
| 58160097602 | NDC | Bexsero vaccine |
| 58160097606 | NDC | Bexsero vaccine |
| 58160097620 | NDC | Bexsero vaccine |

Additional details will be include in the Statistical Analysis Plan (SAP).

#### 9.4. Data Sources

The data for this retrospective secondary data analysis is a large third party payer database, the IQVIA PharMetrics Plus (Pfizer 03 April 2023 version). PharMetrics Plus is a health plan claims database comprised of fully adjudicated medical and pharmacy claims for more than 210 million unique enrollees since 2006. Data contributors to the database are largely commercial health plans. It is representative of the commercially insured US national population for patients under 65 years of age. It contains a longitudinal view of inpatient and outpatient services, prescription and office/outpatient administered drugs, costs, and detailed enrollment information. All data are compliant to the Health Insurance Portability and Accountability Act (HIPAA) to protect patient privacy. The database is used in a variety of life sciences and commercial effectiveness studies. Over 250 peer reviewed publications have used PharMetrics Plus data.

#### 9.5. Study Size

This is an exploratory study, thus no hypothesis was generated. All eligible individuals will be included in the study.

For the sample size estimation, we wished to detect a vaccine effectiveness against gonococcal infection of 20% or more with an onset from 14 days after receipt of both TRUMENBA and MenACWY. A Cox regression of the log hazard ratio on a covariate with a standard deviation of 1.50 to achieve 80% power at a 0.05 significance level to detect a regression coefficient equal to -0.2200, we need a sample of 15,669. The sample size was adjusted for an anticipated overall event rate of 0.0046. We will have 520,392 samples in the study database illustrating that we have adequate samples to conduct the analysis.

#### 9.6. Data Management

This study will use secondary data collected in the PharMetrics Plus database, which is de-identified and HIPAA compliant. The data will be made accessible only to individuals working on the current study. No attempt will be made to identify individual patients, hospitals, or physicians. Analyses will be conducted using Statistical Analysis System (SAS) 9.4 (SAS Institute, Cary, NC).

The analytic files will include person-level data, including information on baseline demographic and clinical characteristics, study outcomes, and vaccination information as described in the variable section above. Data for this study will be processed and managed by Pfizer, Inc., and all analyses will be performed by Pfizer.

#### 9.7. Data Analysis

The zero time is the date of Trumenba vaccination for the exposed group and the date of MenACWY for the unexposed group. We will assess gonococcal infections that occurred between i) 14 days after zero time and 365 days ii) 14 days after zero time and 730 days, iii) 14 days after zero time and 1095 days, and iv) 14 days after zero time and till end of the study period (31Dec2022). We will censor the data in the event of interest, death date (if known), plan disenrollment (if known), target end date, or the end of the study period, whichever comes first. In descriptive analyses, we will fit Kaplan-Meier curves. We will also create unadjusted and covariate adjusted Cox proportional hazard regression models verifying first that the proportionality assumption was satisfied for all independent variables. Hazard ratios (HRs) will be estimated by exponentiation of the coefficient for the vaccine variable in these models, with vaccine effectiveness estimated as (1–HR)×100%. SEs for the coefficients will be used to estimate p values and CIs for the HRs. If a covariate does not satisfy the assumption of proportionality, we will exclude the variable for the multivariable model and will perform the stratified analysis using the covariate.

Detailed methodology for summary and statistical analyses of data collected in this study will be documented in a statistical analysis plan (SAP), which will be dated, filed and maintained by Pfizer. The SAP may modify the plans outlined in the protocol; any major modifications of primary endpoint definitions or their analyses would be reflected in a protocol amendment.

#### 9.8. Quality Control

Only observed data will be used in measuring study variables. It is anticipated that demographic information will be available for nearly all individuals in the study population. All other variables will be defined based on the presence of specific data (eg, diagnosis, procedure, and drug codes) in the analytic file; the absence of such data will be assumed to indicate the absence of the characteristic/event captured by the variable.

#### 9.9. Strengths and Limitations of the Research Methods

#### Strengths

A significant strength of observational retrospective analyses is that they provide a better understanding of the study population in real world clinical practice as compared to the controlled conditions of a clinical trial.

#### Limitations

There are several limitations in this study. Given that this is an observational study using health care administrative claims data, residual confounding due to missing or unmeasured information is possible. To examine this, we will assess the effect of meningococcal vaccination on another sexually transmitted disease occuring, at the same age group, as reference disease outcome. If the HRs in any of these models are less than 1.0, it would indicate that residual confounding exists and may result in adjustment of our vaccine effectiveness (VE) estimates.

Second, health care administrative claims data will be available from 01 January 2016 through 31 December 2022. It is possible that some participants may have received a Trumenba vaccination prior to January 1, 2016 or during a period in which we do not have their claims data and be misclassified as unvaccinated with Trumenba. This may underestimate Trumenba vaccine effectiveness because the Men-ACWY-only cohort will include Trumenba vaccinated patients.

#### 9.10. Other Aspects

Not applicable.

#### 10. PROTECTION OF HUMAN SUBJECTS

#### 10.1. Patient Information

This study involves data that exist in anonymized structured format and contain no patient personal information.

#### 10.2. Patient Consent

As this study involves anonymized structured data, which according to applicable legal requirements do not contain data subject to privacy laws, obtaining informed consent from patients by Pfizer is not required.

#### 10.3. Institutional Review Board (IRB)/Independent Ethics Committee (IEC)

The study databases will be de-identified prior to their release to study investigators, as set forth in the corresponding Data Use Agreement. The study databases have been evaluated and certified by an independent third party to be compliant with the HIPAA of 1996 statistical de-identification standards and to satisfy the conditions set forth in Sections 164.514 (a)-(b)1ii of the HIPAA Privacy Rule regarding the determination and

documentation of statistically de-identified data. Use of the study databases for health services research is therefore fully compliant with the HIPAA Privacy Rule and federal guidance on Public Welfare and the Protection of Human Subjects (45 Code of Federal Regulations [CFR] 46 §46.101) and IRB approval is not required.

#### 10.4. Ethical Conduct of the Study

The study will be conducted in accordance with legal and regulatory requirements, as well as with scientific purpose, value and rigor and follow generally accepted research practices described in Good Pharmacoepidemiology Practices (GPP) issued by the International Society for Pharmacoepidemiology (ISPE), Good Epidemiological Practice (GEP) guidelines issued by the International Epidemiological Association (IEA), Good Outcomes Research Practices issued by the International Society for Pharmacoeconomics and Outcomes Research (ISPOR), International Ethical Guidelines for Epidemiological Research issued by the Council for International Organizations of Medical Sciences (CIOMS), European Medicines Agency (EMA) European Network of Centres for Pharmacoepidemiology and Pharmacoepidemiology, and Food and Drug Administration (FDA) Guidance for Industry: Good Pharmacovigilance and Pharmacoepidemiologic Assessment, and FDA Draft Guidance for Industry and FDA Staff: Best Practices for Conducting and Reporting of Pharmacoepidemiologic Safety Studies Using Electronic Healthcare Data Sets and/or equivalent.

# 11. MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS

This study involves data that exist as structured data by the time of study start.

In these data sources, individual patient data are not retrieved or validated, and it is not possible to link (ie, identify a potential association between) a particular product and medical event for any individual. Thus, the minimum criteria for reporting an adverse event (AE) (ie, identifiable patient, identifiable reporter, a suspect product, and event) cannot be met.

#### 12. PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS

Formal communication of the results of this research will be done by Pfizer authors through peer-reviewed publications. For all publications relating to the Study, Pfizer will comply with recognized ethical standards concerning publications and authorship, including Section II - "Ethical Considerations in the Conduct and Reporting of Research" of the Uniform Requirements for Manuscripts Submitted to Biomedical Journals, http://www.icmje.org/index.html#authorship, established by the International Committee of Medical Journal Editors.

In the event of any prohibition or restriction imposed (eg, clinical hold) by an applicable competent authority in any area of the world, or if party responsible for collecting data from the participant is aware of any new information which might influence the evaluation of the benefits and risks of a Pfizer product, Pfizer should be informed immediately.

#### 13. REFERENCES

- 1. Kuhdari P, Stefanati A, Lupi S, Valente N, Gabutti G. Meningococcal B vaccination: real-world experience and future perspectives. Pathog Glob Health. 2016 Jun-Jul;110(4-5):148-56. doi: 10.1080/20477724.2016.1195072. Epub 2016 Jun 16. PMID: 27309042; PMCID: PMC5072112.
- 2. Wang B, Giles L, Andraweera P, McMillan M, Almond S, Beazley R, Mitchell J, Lally N, Ahoure M, Denehy E, Koehler A, Flood L, Marshall H. Effectiveness and impact of the 4CMenB vaccine against invasive serogroup B meningococcal disease and gonorrhoea in an infant, child, and adolescent programme: an observational cohort and case-control study. Lancet Infect Dis. 2022 Jul;22(7):1011-1020. doi: 10.1016/S1473-3099(21)00754-4. Epub 2022 Apr 12. PMID: 35427492.
- 3. Abara WE, Bernstein KT, Lewis FMT, Schillinger JA, Feemster K, Pathela P, Hariri S, Islam A, Eberhart M, Cheng I, Ternier A, Slutsker JS, Mbaeyi S, Madera R, Kirkcaldy RD. Effectiveness of a serogroup B outer membrane vesicle meningococcal vaccine against gonorrhoea: a retrospective observational study. Lancet Infect Dis. 2022 Jul;22(7):1021-1029. doi: 10.1016/S1473-3099(21)00812-4. Epub 2022 Apr 12. PMID: 35427490.
- 4. Raccagni AR, Galli L, Spagnuolo V, Bruzzesi E, Muccini C, Bossolasco S, Ranzenigo M, Gianotti N, Lolatto R, Castagna A, Nozza S. Meningococcus B Vaccination Effectiveness against Neisseria gonorrhoeae Infection in People Living with HIV: a Case-control Study. Sex Transm Dis. 2023 Jan 13. doi: 10.1097/OLQ.000000000001771. Epub ahead of print. PMID: 36728240.
- 5. Bruxvoort KJ, Lewnard JA, Chen LH, Tseng HF, Chang J, Veltman J, Marrazzo J, Qian L. Prevention of Neisseria gonorrhoeae With Meningococcal B Vaccine: A Matched Cohort Study in Southern California. Clin Infect Dis. 2023 Feb 8;76(3):e1341-e1349. doi: 10.1093/cid/ciac436. Erratum in: Clin Infect Dis. 2023 Jan 11;: PMID: 35642527.
- 6. Abara WE, Bernstein KT, Lewis FMT, Pathela P, Islam A, Eberhart M, Cheng I, Ternier A, Sanderson Slutsker J, Madera R, Kirkcaldy R. Healthy vaccinee bias and MenB-FHbp vaccine effectiveness against gonorrhea. Sex Transm Dis. 2023 Mar 2. doi: 10.1097/OLQ.000000000001793. Epub ahead of print. PMID: 36863060.

#### 14. LIST OF TABLES

- Table 1. Variable List
- Table 2. Diagnosis Codes for Identifying Gonococcal Infections
- Table 3. Diagnosis Codes for Identifying Chlamydial Infections
- Table 4. Current Procedural Terminal Codes and National Drug Codes for Identifying MenACWY Vaccination
- Table 5. Current Procedural Terminal Codes and National Drug Codes for Identifying Trumemba (fHbp) Vaccination
- Table 6. Current Procedural Terminal Codes and National Drug Codes for Identifying Bexsero 4CMenB Vaccination

#### 15. LIST OF FIGURES

None.

#### ANNEX 1. LIST OF STAND ALONE DOCUMENTS

None.

## **Document Approval Record**

**Document Name:** B1971066\_Non Interventional Study Protocol\_18April2023

**Document Title:** B1971066\_Non Interventional Study Protocol\_18April2023

| Signed By: | Date(GMT) | Signing Capacity |
|------------|----------------------|------------------------|
| PPD | 19-Apr-2023 19:31:05 | Business Line Approver |
| | 19-Apr-2023 21:52:10 | Author Approval |
| | 21-Apr-2023 16:33:13 | Scientific Review |